CLINICAL TRIAL: NCT01484418
Title: Exposure Therapy in Chronic Low Back Pain Patients
Brief Title: Exposure-based Treatment for Avoidant Back Pain Patients
Acronym: ETABP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other); German Research Foundation (Other)
Responsible Party: Principal Investigator, Julia Anna Glombiewski, Ph.D, Licensed Psychologist, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFG-GL 607
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Cognitive Behavioural Therapy; Exposure; Fear avoidance; Cognitive Behavioural Therapy in chronic low back pain; Exposure in vivo in chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A Exposure long (Experimental): Exposure in vivo for fear avoidant chronic low back pain patients. This treatment means that the individual is exposed to movements and tasks that have been avoided due to fear of (re)injury. The treatment begins after three educational lessons including the rational and developing a fear hierarchy. Exposure phase includes 10 exposures sessions which are highly individualized. Behavioral experiments can be included to correct catastrophic misinterpretations. The main purpose of this intervention type is to reduce pain related disability via diminishing fear avoidance.
  Interventions: Behavioral: Exposure in vivo
- B Exposure short (Experimental): See above exposure long. This treatment comprises 5 exposure sessions.
  Interventions: Behavioral: Exposure in vivo
- C Cognitive behavioural psychotherapy (Active Comparator): Cognitive behavioural psychotherapy for fear avoidant chronic low back patients. The therapy is modularized in three main parts. The educational lesson is followed by the module graded activity which represents the behavioral part of the program. The second module comprises relaxation. And the last part contains cognitive interventions. Cognitive behavioural intervention techniques are employed to support the patient in the process of coping with chronic pain: i.e. reduction of disability and improving functional ability.
  Interventions: Behavioral: Cognitive Behavioural Psychotherapy

INTERVENTIONS:
Behavioral: Exposure in vivo — 5-10 sessions based on an individualized fear hierarchy
  Arms: A Exposure long; B Exposure short
Behavioral: Cognitive Behavioural Psychotherapy — graded activity, relaxation techniques and cognitive interventions
  Arms: C Cognitive behavioural psychotherapy

SUMMARY:
Chronic low back pain often results in psychosocial and physical disability. A subgroup of these patients shows fear of (re)injury and avoidance behaviour leading to higher disability. The purpose of this study is to determine whether exposure in vivo is more effective in the treatment of fear avoidant chronic back pain patients than psychological treatment as usual (cognitive behavioural psychotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Having at least 3 months back pain
* Sufficient level on fear avoidance scores (TSK, Phoda)
* Being German-speaking
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* Red flags
* Pregnancy
* Illiteracy
* Psychoses
* Alcohol addiction
* surgeries during the last 6 months or planed surgeries
* Specific medical disorders or cardiovascular diseases preventing participation in physical exercise
* Participating in another psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain severity at 3 and 6 months after admission | from Pretest (admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Numeric Rating Scale (NRS)
Change from baseline in pain disability at 3 and 6 months after admission | from Pretest (admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Pain Disability Index (PDI) Quebec Back Pain Disability Scale (QBPDS)

SECONDARY OUTCOMES:
Change in fear avoidance from Pretest to two in-between time points to Posttest | from Pretest (admission) to one in-between timepoint (an expected 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Tampa Scale of Kinesiophobia (TSK) Pain Anxiety Symptom Scale (PASS)
Change in pain catastrophizing from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to one in-between timepoint (an expected 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Pain Catastrophizing Scale (PCS)
Change in emotional distress from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to one in-between timepoint (an expected 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Hospital Anxiety and Depression Scale (HADS)
Change in quality of life from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to one in-between timepoint (an expected 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  EuroQol (EQ-5D)
Change in physical activity from Pretest to two in-between timepoints to Posttest to Follow-up Time | from Pretest (admission) to one in-between timepoint (an expected 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  International Physical Activity Questionnaire(IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof., Study Director — Philipps University Marburg, Department of Clinical Psychology and Psychotherapy; Julia A. Glombiewski, Dr., Study Chair — Philipps University Marburg, Department of Clinical Psychology and Psychotherapy
Locations (1):
- Philipps University Marburg, Department of Clinical Psychology and Psychotherapy, Marburg, Germany

REFERENCES:
- [Derived] Glombiewski JA, Holzapfel S, Riecke J, Vlaeyen JWS, de Jong J, Lemmer G, Rief W. Exposure and CBT for chronic back pain: An RCT on differential efficacy and optimal length of treatment. J Consult Clin Psychol. 2018 Jun;86(6):533-545. doi: 10.1037/ccp0000298. PMID 29781651
- [Derived] Riecke J, Holzapfel S, Rief W, Glombiewski JA. Evaluation and implementation of graded in vivo exposure for chronic low back pain in a German outpatient setting: a study protocol of a randomized controlled trial. Trials. 2013 Jul 9;14:203. doi: 10.1186/1745-6215-14-203. PMID 23837551
- See also: Related Info — http://www.uni-marburg.de/fb04/ag-klin/mitarbeiter/jglombiewski